CLINICAL TRIAL: NCT06645314
Title: Study on the Safety and Efficacy of BST06 Injection in the Treatment of Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Collaborators: South China Hospital of Shenzhen University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BST06-001
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BST06 (Experimental): intravenous infusion
  Interventions: Biological: Group A; Biological: Group B

INTERVENTIONS:
Biological: Group A — 3.0 × 10 ^ 9 BST06 cells, intravenous infusion，at least 2 subjects enrolled, up to a maximum of 8 subjects enrolled
Biological: Group B — 3.0 × 10 ^ 10 BST06 cells, intravenous infusion, at least 2 subjects enrolled, up to a maximum of 8 subjects enrolled

SUMMARY:
The study is an exploratory clinical trial initiated by an open, single arm researcher to evaluate the safety, tolerability, and preliminary efficacy of BST06 injection in the treatment of advanced hepatocellular carcinoma in subjects. This study plans to apply Bayesian Optimal Interval (BOIN) design, with at least 2 and up to 8 DLT assessable subjects in each dose group, who must complete a 28 day DLT assessment period. The study plan includes 2 dose groups: 5x10 ^ 9 and 3x10 ^ 10 BST06 cells

DETAILED DESCRIPTION:
Main purpose:

Evaluate the safety and tolerability of BST06 injection in the treatment of advanced hepatocellular carcinoma in subjects.

Secondary purpose:

1. Evaluate the preliminary effectiveness of BST06 injection in the treatment of advanced hepatocellular carcinoma in subjects:
2. Evaluate the pharmacokinetic (PK) characteristics of BST06 injection.

Exploratory purpose:

Explore the Pharmacodynamics (PD) characteristics of BST06 injection.

ELIGIBILITY:
Inclusion Criteria:

* 1: The age range is 18-70 years old (including the critical value);
* 2: HCC patients diagnosed by histopathological or cytological examination, or those who meet the criteria of the American Association for the Study of the Liver (AASLD) or are clinically diagnosed with hepatocellular carcinoma according to the "2022 Guidelines for the Diagnosis and Treatment of Primary Liver Cancer";
* 3: Tumor tissue pathology immunohistochemistry GPC3 positive;
* 4: Patients who have undergone at least first-line systemic therapy and have experienced disease progression confirmed by imaging (including but not limited to systemic chemotherapy, targeted therapy, immunotherapy, etc.), have been evaluated by the researchers to have refused other standard treatments at the time of enrollment, or have been determined by the researchers to have difficulty benefiting from treatments recommended by domestic and foreign clinical guidelines or expert consensus.
* 5: At least one tumor lesion has not received radiation therapy or other local treatments within 28 days. Moreover, according to the researchers' judgment, at least 2 intact tumor puncture samples with a length of ≥ 2cm can be obtained through surgical resection or puncture, which can be from different lesions, for the preparation of BST06 cells;
* 6: After TIL sampling, there should be at least one measurable lesion that meets the mRECIST standard definition (RECIST 1.1 standard for subjects without intrahepatic lesions);
* 7: Eastern Cooperative Oncology Group (ECOG) score ≤ 1 point;
* 8: Child Pugh liver function grading score A-B7
* 9: HBsAg positive patients must meet the requirement of HBV DNA quantification<1 * 104 IU/ml (or 5 * 104 copy/ml) or receive at least one week of anti HBV treatment with a 10 fold reduction in viral index before the start of the study
* 10: Expected survival time ≥ 3 months;
* 11: During the screening and preparation period (within 14 days prior to TIL sampling), sufficient organ and bone marrow function was assessed
* 12: Prior to TIL sampling, adverse reactions caused by previous treatments had already recovered to the Common Adverse Event Evaluation Criteria (CTCAE) of 5.0 ≤ 2 (excluding toxicity judged by researchers to have no safety risk, such as hair loss or peripheral neurotoxicity of grade 2 or below);
* 13: From signing the informed consent form to agreeing to take effective contraceptive measures within 6 months after BST06 cell transfusion (subjects must use non pharmacological contraception);
* 14: Those who fully understand this experiment and voluntarily sign the informed consent form, and are able to comply with the visit and related procedures specified in the protocol.

Exclusion Criteria:

* 1: Pregnant or lactating women;
* 2: Subjects with a history of severe allergies and allergies to experimental drugs including but not limited to cyclophosphamide, fludarabine, BST06 injection components, etc;
* 3: Past or current presence of hepatic encephalopathy; Known patients with untreated or uncontrolled central nervous system metastases; Except for those who have received treatment and have stable symptoms, and have stopped glucocorticoid and anticonvulsant drug treatment for ≥ 4 weeks before pre-treatment;
* 4: At present, clinically significant ascites exists, defined as ascites with positive physical examination signs or requiring intervention treatment control (only those with imaging showing ascites without intervention can be included);
* 5: The proportion of liver tumors is ≥ 50%. For subjects planning to undergo liver lesion resection for specimen collection and preparation, the indocyanine green 15 minute retention rate (ICG-R15) must be ≥ 30%;
* 6: Organ transplantation, history of hematopoietic stem cell transplantation;
* 7: Other serious diseases that may restrict participants from participating in this trial;
* 8: HIV positive, or positive for Treponema pallidum antibody; For patients with active hepatitis B or C, it is recommended to continue taking antiviral drugs during the study period. Active hepatitis B is defined as: positive hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg), and HBV-DNA>10000 IU/ml. Active hepatitis C is defined as HCV RNA above the lower limit of detection;
* 9: Within the 4 weeks prior to TIL sampling, any immunosuppressive drugs such as corticosteroids were used, or it was determined by the researcher that there were comorbidities that required the use of immunosuppressive drugs during the trial period. But it is allowed to use physiological doses of glucocorticoids (i.e. not exceeding 15mg/day of prednisone or equivalent doses of other glucocorticoids), and inhaled, intranasal, topical, or prophylactic corticosteroids are allowed to be used for contrast agent allergies;
* 10: Received local treatments such as interventional therapy, radiotherapy, ablation, as well as systemic treatments (including small molecule targeting, anti-PD-1/PD-L1 monoclonal antibodies, and chemotherapy) within 4 weeks prior to pre-treatment. Or received thymosin, interferon and other immunotherapy or any Chinese herbal medicine or traditional Chinese patent medicines and simple preparations for tumor control within 1 week before pretreatment;
* 11: Individuals who have received a live vaccine within the first 3 months of screening or plan to receive a live vaccine during the trial period
* 12: Individuals who have undergone major surgery (≥ grade 3 surgery) within the 4 weeks prior to screening, or who require elective surgery during the trial period (excluding TIL sampling surgery);
* 13: Patients who experience surgical complications or delayed wound healing prior to pre-treatment, and who have been assessed by researchers to increase the risk of gonorrhea, TIL treatment, or infection;
* 14: Diagnosed within 5 years prior to screening as coexisting with other primary malignant tumors, excluding skin basal cell carcinoma, skin squamous cell carcinoma, and/or carcinoma in situ that has undergone radical resection;
* 15: Received cell therapy products within 6 months prior to pre-treatment;
* 16: Known cases of alcohol abuse, drug use, or substance abuse, as well as those deemed unsuitable by other researchers to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | From the infusion (Day 0) to Day 28
  DLT is defined as the following adverse events related to the investigational drug(definitely related, likely related,possibly related) that occur within 28 days after administration of BST08 (using CTCAE 5.0 or CRS grading criteria): (1) hematological toxicity; (2) Grade 3 non hematological toxicity lasting for more than 7 days, or ≥ Grade4 non hematological toxicity, regardless of duration, but excluding the following situations; (3)Cytokine Release Syndrome(CRS)
Maximum ToleratedDose(MTD) | From the infusion (Day 0) to Day 28
  The highest dose of DLT observed in subjects with less than 2/6 (at least 6 subjects in this experimental group received BST08 administration and completed DLT observation)

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Han, PhD, Principal Investigator — South China Hospital of Shenzhen Univercity; Yuqing Li, PhD, Principal Investigator — South China Hospital of Shenzhen Univercity